CLINICAL TRIAL: NCT03049358
Title: Olfactory Training For Post Radiation Olfactory Loss In Patients With Paranasal Sinus and Nasopharyngeal Carcinoma
Brief Title: Olfactory Training in Improving Sense of Smell After Radiation Therapy in Patients With Paranasal Sinus or Nasopharyngeal Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Accrual factor
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: ENT0059; NCI-2017-00147 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); IRB-39817 (Other: Stanford IRB)
Record Dates: First submitted 2017-02-06; First posted 2017-02-10 (Actual); Last update posted 2019-02-05 (Actual); Status verified 2019-02

CONDITIONS: Stage 0 Nasopharyngeal Carcinoma; Stage 0 Paranasal Sinus Cancer; Stage I Nasopharyngeal Carcinoma; Stage I Paranasal Sinus Cancer; Stage II Nasopharyngeal Carcinoma; Stage II Paranasal Sinus Cancer; Stage IIA Nasopharyngeal Carcinoma; Stage IIB Nasopharyngeal Carcinoma; Stage III Nasopharyngeal Carcinoma; Stage III Paranasal Sinus Cancer; Stage IV Nasopharyngeal Carcinoma; Stage IV Paranasal Sinus Cancer; Stage IVA Nasopharyngeal Carcinoma; Stage IVA Paranasal Sinus Cancer; Stage IVB Nasopharyngeal Carcinoma; Stage IVB Paranasal Sinus Cancer; Stage IVC Nasopharyngeal Carcinoma; Stage IVC Paranasal Sinus Cancer
MeSH Terms: conditions — Nasopharyngeal Carcinoma; Paranasal Sinus Neoplasms | interventions — Coal Tar; Therapeutics; Eucalyptus Oil

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm I (olfactory training) (Experimental): Patients undergo olfactory training by smelling 4 essential oils in vials (rose, lemon, clove, and eucalyptus) over 15 seconds each, twice daily for 12 weeks.
  Interventions: Other: Physiologic Testing; Other: Quality-of-Life Assessment; Procedure: Therapeutic Procedure; Other: rose essential oil; Other: lemon essential oil; Other: clove essential oil; Other: eucalyptus essential oil
- Arm II (sham training) (Sham Comparator): Patients undergo sham training by smelling canola oil in 4 vials over 15 seconds each, twice daily for 12 weeks.
  Interventions: Other: Physiologic Testing; Other: Quality-of-Life Assessment; Procedure: Sham Intervention; Other: canola oil placebo

INTERVENTIONS:
Other: Physiologic Testing — Undergo UPSIT smell test
  Other Names: Physiologic Test; Study of Physiologic Variables
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Procedure: Sham Intervention — Undergo sham training
  Arms: Arm II (sham training)
Procedure: Therapeutic Procedure — Undergo olfactory training
  Other Names: Therapeutic Interventions; Therapeutic Method; Therapeutic Technique; Therapy; TREAT; Treatment
  Arms: Arm I (olfactory training)
Other: rose essential oil — patient smells rose oil in vial
  Arms: Arm I (olfactory training)
Other: lemon essential oil — patient smells lemon oil in vial
  Arms: Arm I (olfactory training)
Other: clove essential oil — patient smells clove oil in vial
  Arms: Arm I (olfactory training)
Other: eucalyptus essential oil — patient smells eucalyptus oil in vial
  Arms: Arm I (olfactory training)
Other: canola oil placebo — patient smells canola oil in vial
  Arms: Arm II (sham training)

SUMMARY:
This randomized phase I trial studies how well olfactory training works in improving sense of smell after radiation therapy in patients with paranasal sinus or nasopharyngeal cancer. Olfactory training may improve smell function after radiation therapy in patients with paranasal sinus or nasopharyngeal cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the effect of olfactory training on olfactory function in patients with paranasal sinus and nasopharyngeal carcinoma suffering from olfactory loss after radiation.

SECONDARY OBJECTIVES:

I. To evaluate the possible effect of olfactory training on quality of life in patients with paranasal sinus and nasopharyngeal carcinoma suffering from olfactory loss after radiation.

II. To study rate and severity of olfactory dysfunction after radiation therapy in patients with paranasal sinus or nasopharyngeal carcinoma.

III. To evaluate the possible preventive effect of olfactory training on olfactory dysfunction in patients with paranasal sinus and nasopharyngeal carcinoma who will undergo radiation therapy.

OUTLINE: Patients are randomized to 1 of 2 arms. Arm I: Patients undergo olfactory training by smelling 4 essential oils in vials (rose, lemon, clove, and eucalyptus) over 15 seconds each, twice daily for 12 weeks.

Arm II: Patients undergo sham training by smelling canola oil in 4 vials over 15 seconds each, twice daily for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Eligible disease(s)/stage(s): nasopharyngeal carcinoma, paranasal sinus cancers/any stage
* Patients with paranasal sinus or nasopharyngeal carcinoma who are about to undergo radiation therapy; patients with paranasal sinus or nasopharyngeal carcinoma who have completed radiation therapy 3-6 months prior to enrollment who then show olfactory loss on a screening test (University of Pennsylvania Smell Identification Test [UPSIT] - score of 34 or 33 or lower out of 40, depending on female/male); both those patients undergoing chemotherapy and those who did not will be eligible, and this factor will be assessed as a possible confounder/contributor in a multi-regression analysis
* No race-ethnic restriction
* No life expectancy restriction
* No need for Karnofsky performance status
* Only requirement for organ function is for patients to have competency to consent and participate in the study; in the arm of the study which requires patients to have olfactory dysfunction before enrollment, an UPSIT score will be used to identify these patients
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* No therapy restrictions
* No restrictions on use of other investigational agents
* Co-morbid disease or incurrent illness such as:

  * History of head trauma
  * History of nasal surgery other than biopsy (before cancer was diagnosed)
  * History of sinus surgery other than biopsy (before cancer was diagnosed)
  * Chronic rhinosinusitis with or without polyp
  * Pregnancy
  * Cognitive dysfunction
  * History of brain surgery
  * Psychiatric or neurologic diseases interfering with sense of smell
  * Congenital disorders of olfactory dysfunction
  * Olfactory loss prior to onset of nasopharyngeal carcinoma
* No allergic reactivity has been associated with olfactory training and thus there is no need for any exclusion criteria related to this
* No other agents have any possible potentiation or decreased activity related to olfactory training and thus there is no need for any exclusion criteria related to this
* There are no other agent-specific exclusion criteria
* Pregnant women will be excluded; nursing patients will be included

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2018-10 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
Change in olfactory function in patients with paranasal sinus or nasopharyngeal carcinoma after completion of radiation therapy as measured by UPSIT score | Baseline to 12 weeks
  T-test or Mann-Whitney U test, where appropriate, will be used for comparing continuous variables, and chi-squared test will be used for comparing categorical variables. Continuous UPSIT score will be summarized using the following statistics: number of subjects, arithmetic mean, standard deviation, median, first quartile, third quartile, minimum, and maximum values. The dependent variable UPSIT score will be either the percent change from baseline or change from baseline in the endpoint. Mixed model repeated measures (MMRM) analysis will be used and the model will included fixed effect terms

SECONDARY OUTCOMES:
Efficacy of olfactory training during radiation therapy as measured by change in UPSIT scores | Baseline
  T-test or Mann-Whitney U test, where appropriate, will be used for comparing continuous variables, and chi-squared test will be used for comparing categorical variables. Continuous UPSIT score will be summarized using the following statistics: number of subjects, arithmetic mean, standard deviation, median, first quartile, third quartile, minimum, and maximum values. The dependent variable UPSIT score will be either the percent change from baseline or change from baseline in the endpoint. Mixed model repeated measures (MMRM) analysis will be used and the model will included fixed effect terms
Improvement in quality of life related to olfactory dysfunction as measured by change in the Questionnaire of Olfactory Disorders (QOD) score | Baseline to 12 weeks
  Within each subgroup of participants, change in QOD score after olfactory training will be calculated and compared between treatment and control group. Confidence interval (CI) 95% and P value < 5% will be set as statistical parameters to define if noted difference is significant. Based on previous studies, a change of >= 1/2 standard deviation of the pre-treatment score would be clinically significant.
Severity of olfactory dysfunction after completion of radiation therapy as measured by UPSIT score | Baseline
  T-test or Mann-Whitney U test, where appropriate, will be used for comparing continuous variables, and chi-squared test will be used for comparing categorical variables. Continuous UPSIT score will be summarized using the following statistics: number of subjects, arithmetic mean, standard deviation, median, first quartile, third quartile, minimum, and maximum values. Continuous UPSIT score will be summarized using the following statistics: number of subjects, arithmetic mean, standard deviation, median, first quartile, third quartile, minimum, and maximum values. These statistics will be shown

CONTACTS AND LOCATIONS:
Overall Officials: Zara Patel, Principal Investigator — Stanford University
Locations (1):
- Stanford University, School of Medicine, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No